CLINICAL TRIAL: NCT06432439
Title: Microneedling And Its Effect On Outcome Of Root Coverage With Coronally Advanced Flap Involving Isolated RT1 Maxillary Gingival Recession In Thin Gingival Phenotype: A Randomized Controlled Clinical Trial
Brief Title: Impact of Microneedling on Coverage of RT1 Gingival Recession in Thin Phenotype.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Amisha perio
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Gingival Recession, Localized
Keywords: microneedling; phenotype; gingival recession; coronally advanced flap
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEST GROUP (Experimental): Isolated RT1 gingival recession treated by microneedling followed by Coronally Advanced Flap procedures
  Interventions: Procedure: microneedling followed by CAF procedures
- CONTROL GROUP (Active Comparator): Isolated RT1 gingival recession treated by Coronally Advanced Flap procedures alone.
  Interventions: Procedure: CAF procedure

INTERVENTIONS:
Procedure: microneedling followed by CAF procedures — microneedling will be done on gingiva of RT1 recession tooth in 4 sessions followed by CAF 2months later for root coverage
  Arms: TEST GROUP
Procedure: CAF procedure — RT1 gingival recession coverage by CAF procedures alone.
  Arms: CONTROL GROUP

SUMMARY:
Gingival Recession (GR) is a common finding in among adults, regardless of the oral hygiene levels. When it is associated with esthetic impairment, dentin hypersensitivity, root caries, surgical treatment is indicated. Mid-buccal Gingival Recessions are an extremely prevalent condition and have root coverage potential through periodontal plastic surgery procedures.

A flap thickness of > 0.8 mm results in a covered root surface of 100%, whereas a flap thickness of < 0.8 mm results in partial root coverage in Coronally Advanced Flap (CAF)procedure.

The present study aims to increase the gingival thickness by microneedling procedures to enhance root coverage by CAF procedures in thin gingival phenotype.

DETAILED DESCRIPTION:
Gingival recession is defined as the migration of the marginal tissue toward the apical of the cementoenamel junction. It is one of the most common mucogingival deformities requiring surgical correction. The rationale for treating buccal recessions are mainly aesthetic concerns, and clinical situations where unfavourable contour of the gingival margin might be an obstacle for proper plaque control. Cairo et al in 2018 categorised GRs into 3 types with reference to interdental clinical attachment loss as RT1, RT2 and RT3. Mid-buccal GRs have root coverage potential through periodontal plastic surgery procedures. Coronally positioned flap is a simple and predictable treatment of gingival recession defects. It has been observed that a flap thickness of > 0.8 mm results in a covered root surface of 100%, whereas a flap thickness of < 0.8 mm results in partial root coverage in CAF procedure. Microneedling (MN), creates microinjuries that result in minimal superficial bleedings and create a wound-healing cascade from which various growth factors are released. MN as opposed to Connective Tissue Grafts is a non-surgical approach to increase gingival thickness, that results in significant changes in the Gingival Thickness of individuals with thin gingival phenotype.

ELIGIBILITY:
INCLUSION CRITERIA:

* Presence of isolated (RT1) by Cairo et al 2011 buccal maxillary gingival recessions in esthetic zone including maxillary central incisors, lateral incisors and canines associated with esthetic complaints and/or dental sensitivity and otherwise systemically healthy.
* Gingival Recession ≥2mm and clinically identifiable CEJ
* Age 20years-50 years
* Patient demonstrating compliance for maintaining good oral hygiene after Phase 1 thearpy Plaque index (PI) <1, Gingival Index (GI) <1
* Providing a written and verbal informed consent.

EXCLUSION CRITERIA

* Patient with systemic disease that can influence the outcome of therapy.
* Pregnant females or on oral contraceptive pills or hormone replacement therapy.
* Smokers and patients undergoing orthodontic therapy
* Physically and mentally impaired patients.
* Non vital, malpositioned tooth
* Presence of cervical abrasions or restorations in the area
* Previous history of periodontal surgery on the involved sites.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recession Depth | 3 months
  recorded in mm with a periodontal probe from the cementoenamel junction to the crest of the gingival margin at mid labial region.
RECESSION WIDTH (RW) | 3 months
  recorded in mm with a periodontal probe from the mesial to distal gingival margin at the level of cementoenamel junction.
ROOT COVERAGE PERCENTAGE | 3 months
  calculated according to the formula Root Coverage percentage = Recession depth (preop-postop)*100 Recession depth preoperative
Gingival thickness(GT) | 3 months
  GT is measured with the help of No:15 endodontic spreaders with silicon disc as stopper was inserted perpendicularly at 1.5mm apical to gingival margin, till the hard tissue was felt. The depth of penetration was noted using digital calliper

SECONDARY OUTCOMES:
CLINICAL ATTACHMENT LEVEL (CAL) | 3 months
  Clinical attachment level will be measured as the distance between the cemento- enamel junction and the base of pocket. Measurements will be made at 6 sites of each tooth
Probing Pocket Depth (PPD) | 3 months
  Probing pocket depth will be measured as the distance from gingival margin to the base of pocket. The probing depth measurements will be assessed using the Periodontal probe
Bleeding on Probing (BOP) | 3 months
  It will be measured by walking the periodontal probe at 6 sites of each tooth
Plaque Index (PI) | 3 months
  For the scoring, a mouth mirror, an explorer and a light source will be used on air dried teeth and gingiva
Gingival Index (GI | 3 months
  Gingival index by Loe and Silness (1963)22 will be used to assess severity of gingival inflammation
Keratinized Tissue Width (KTW) | 3 months
  Keratinized tissue width will be measured with the help of UNC 15 probe with silicon stopper from the mucogingival junction to the free gingival margin and measured on vernier caliper

CONTACTS AND LOCATIONS:
Overall Officials: Amisha Goyal, BDS, Principal Investigator — PGIDS